CLINICAL TRIAL: NCT04771156
Title: Ketorolac in Palatoplasty: A Randomized Blinded Controlled Trial.
Brief Title: Ketorolac in Palatoplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Matthew Greives, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-21-0044
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Ketorolac) (Experimental)
  Interventions: Drug: Ketorolac
- Control Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — Ketorolac 0.5mg/kg will be administered intra-operatively at the conclusion of the case and 3 more doses scheduled every 8 hours in the first 24 hours post-operatively for a total of 4 doses of Ketorolac
  Arms: Experimental group (Ketorolac)
Drug: Placebo — 0.9% Normal Saline will be administered intra-operatively at the conclusion of the case and 3 more doses scheduled every 8 hours in the first 24 hours post-operatively for a total of 4 doses of normal saline.
  Arms: Control Group

SUMMARY:
The purpose of this study is to see if the addition of IV Ketorolac to usual care multi-modal pain therapy compared to usual care will improve oral intake post-operatively

ELIGIBILITY:
Inclusion Criteria:

-Patient with Cleft palate (Complete and incomplete), with or without cleft lip, unilateral or bilateral

Exclusion Criteria:

* Syndromic Cleft Palate patients
* Previous palatoplasty
* Major unrepaired cardiac malformation
* History of GI complications (GI Bleed, Gastric Ulceration)
* History of Renal disorder
* History of coagulopathy (As contraindication to NSAID use)
* Feeding tube dependency
* Patients whose parents refuse to consent to randomization

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Volume of oral intake | from arrival to Post-Anesthesia Care Unit (PACU) to 24 hours post surgery
  This will be measured in mL's of fluids

SECONDARY OUTCOMES:
Pain as assessed by the Faces, Legs, Activity, Cry, Consolability (FLACC) scale | immediately upon arrival at PACU
  This scale has 5 questions and each is scored from 0-2,higher number indicating a worse outcome
Pain as assessed by the Faces, Legs, Activity, Cry, Consolability (FLACC) scale | 24 hours post surgery
  This scale has 5 questions and each is scored from 0-2,higher number indicating a worse outcome
Pain as assessed by the Faces, Legs, Activity, Cry, Consolability (FLACC) scale | 48 hours post surgery
  This scale has 5 questions and each is scored from 0-2,higher number indicating a worse outcome
Pain as assessed by the Faces scale | 7 days post discharge
  Subjective assessment of discomfort by parent, scored from 1-10, higher number indicating a worse outcome
Time to first oral intake | within 24 hours post surgery
Number of participants with Post-operative bleeding that requires either transfusion or Unplanned return to Operating Room | 24 hours and 48 hours after surgery
Amount of Post-operative narcotic usage (recorded in Morphine milligram Equivalents) | 7 days post surgery
Number of participants who need narcotic prescription at discharge | at discharge(24-48 hours post surgery)
Renal function measured in mL/kg of urine output | from arrival to PACU to discharge (24-48 hours post surgery)
Number of participants with post operative complications | 30 days post surgery
  post operative complications include,Unplanned return to OR, ER or unplanned clinic visit , Infection, Fever

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Grieves, MD,MS,FACS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No